CLINICAL TRIAL: NCT05405335
Title: Effect of Prone Positioning on the Severity of COVID-19 Pneumonia and Acute Respiratory Distress Syndrome. A Randomized Clinical Trial
Brief Title: Effect of Prone Positioning on the Severity of COVID-19 Pneumonia and Acute Respiratory Distress Syndrome.
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayub Medical College, Abbottabad (Other)
Collaborators: Ayub Teaching Hospital (Other)
Responsible Party: Principal Investigator, Hamza Javed, Doctor, Ayub Medical College, Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AyubMC
Record Dates: First submitted 2022-06-02; First posted 2022-06-06 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; COVID-19 Pneumonia; Prone Positioning
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: parallel groups randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Positioned Group (Experimental): Intermittent prone positioning for a total of eight hours per day for seven days. Each cycle of prone positioning should not be less than 30 minutes and note more than 3 hours at one time.
  Rest of the treatment as per protocols of the institution
  Interventions: Other: Prone Positioning Maneuver
- Control Group (No Intervention): Treatment as per institutional protocols- the protocols does not involve prone positioning of the patients

INTERVENTIONS:
Other: Prone Positioning Maneuver — intermittent prone positioning for eight hours per day for seven days. each cycle should not be less than 30 minutes or more than 3 hours.
  Other Names: Prone Positioning
  Arms: Prone Positioned Group

SUMMARY:
With this research, we are aiming at finding out the effectiveness of prone positioning in this region population affected by moderate pneumonia due to covid 19 infection so that the hospital staff and doctors may be encouraged with facts and data to use such an easy maneuver to stabilize patient's oxygen saturation as we believe that prone positioning does have a protective effect against severe disease and has an effect on reducing mortality if patients are encouraged for prone positioning with proper technique and for suitable time duration as has been observed in the clinical practice in the covid wards. Therefore, we want to assess the effects of 8 hours per day prone positioning the patients with confirmed covid pneumonia admitted in the covid wards.

DETAILED DESCRIPTION:
Currently, Pakistan and specifically the Hazara division is being badly hit by the fourth wave of covid 19. Patients are mostly presenting with covid pneumonia with or without other complications such as ARDS, ARF, and shock. A nationwide vaccination drive has been launched in collaboration with the WHO but the general population's response towards getting self-vaccinated is not very much appreciable.

It has been reported in a study from new jersey that awake prone positioning in a spontaneously breathing patients can improve arterial blood oxygen saturation.1 another systematic review of 50 articles, including a total of 2994 patients among which 921 patients were managed with awake prone positioning and the rest by usual care, reported significant improvement in oxygenation parameters with prone positioning. They also concluded that it did not reduce the invasive ventilation rate. 2 another meta-analysis of randomized controlled trials suggested that prone positioning has a protective effect on the lungs by improving oxygenation and can reduce mortality in patients with acute respiratory distress syndrome (ARDS) but also suggested further investigations through randomized clinical trials into the effectiveness of prone positioning in covid 19 associated ARDS. 3

In a report of original investigations, K Solverson et al. concluded that prolonged prone positioning improved oxygenation parameters and reduce mortality but the patients could not tolerate such a long duration. They also suggested a further investigation into the methods to improve the tolerability of awake prone positioning and its long-term benefits.4 Gattinoni L et al. in their multisystem randomized clinical trial where they prone positioned patients for 6 hours per day for a period of 10 days reported that it does improve the oxygenation but it does not improve survival.5 In a randomized controlled trial, Taccone P, reported similar 28th-day and 6th-month outcomes in patients with moderate and severe hypoxemia.6 similar results were reported by Martha A. Q. Curley et al in their study on the pediatric population.7 Guerin C et al. reported no beneficial effects on survival although they did conclude that prone positioning has a protective effect against ventilator-associated pneumonia.8 Ehrmann S et al. in their randomized, controlled, multinational, open-label meta-trial, reported that awake prone positioning of patients with hypoxaemic respiratory failure due to COVID-19 reduces the incidence of treatment failure and the need for intubation without any signal of harm. Their results support the routine use of the prone positioning technique in patients with COVID-19. 9 Binda F et al. in their cross-sectional study on the complications related to prone positioning although considered safe and feasible but reported the prevalence of many complications associated with prone positioning such as pressure ulcers, bleeding from the upper airways, and medical device displacement.10. Malik GR et al. also reported some peripheral nerve injuries especially in the arms after their experience with prone positioning of patients in four tertiary care hospitals.11 None of these complications are immediately fatal and can be managed easily while the patients are in the hospital.

With this research, we are aiming at finding out the effectiveness of prone positioning in this region population affected by moderate pneumonia due to covid 19 infection so that the hospital staff and doctors may be encouraged with facts and data to use such an easy maneuver to stabilize patient's oxygen saturation as we believe that prone positioning does have a protective effect against severe disease and has an effect on reducing mortality if patients are encouraged for prone positioning with proper technique and form suitable time duration as has been observed in the clinical practice in the covid wards. Therefore, we want to assess the effects of 8 hours per day prone positioning the patients with confirmed moderately severe covid pneumonia admitted in the covid wards.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed covid pneumonia/ acute respiratory distress syndrome cases

Exclusion Criteria:

* consent denial, patients having contraindications to prone positioning such as shock, acute bleeding, trauma, spinal instability, raised Intracranial Pressure, sternal/ tracheal surgery, Female pregnant patients in 2nd and 3rd trimester

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
percentage of patients dying COVID-19 pneumonia/ ARDS in both groups | Three months
  Effect of prone positioning on the mortality of patients suffering from covid pneumonia/ acute respiratory distress syndrome

SECONDARY OUTCOMES:
Respiratory physiology- mean PaO2 and Mean respiratory rate of both groups at first, seventh and fiourteenth day of admission | Three months
  effects on the PaO2, respiratory rate and mask type (supplemental oxygen requirement)

CONTACTS AND LOCATIONS:
Overall Officials: Hamza Javed, MBBS, Principal Investigator — Ayub Teaching Hospital, ABbottabad
Locations (1):
- Ayub Teaching Hospital, Abbottābād, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson SA, Horton DJ, Fuller MJ, Yee J, Aliyev N, Boltax JP, Chambers JH, Lanspa MJ. Patient-directed Prone Positioning in Awake Patients with COVID-19 Requiring Hospitalization (PAPR). Ann Am Thorac Soc. 2021 Aug;18(8):1424-1426. doi: 10.1513/AnnalsATS.202011-1466RL. No abstract available. PMID 33596394
- [Background] Oliveira VM, Weschenfelder ME, Deponti G, Condessa R, Loss SH, Bairros PM, Hochegger T, Daroncho R, Rubin B, Chiste M, Batista DC, Bassegio DM, Nauer Wda S, Piekala DM, Minossi SD, Santos VF, Victorino J, Vieira SR. Good practices for prone positioning at the bedside: Construction of a care protocol. Rev Assoc Med Bras (1992). 2016 May-Jun;62(3):287-93. doi: 10.1590/1806-9282.62.03.287. PMID 27310555

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT05405335/Prot_SAP_ICF_001.pdf